CLINICAL TRIAL: NCT05045573
Title: Pathological Results After Downstaging of Agressive Hepatocellular Carcinoma Using 90Y-SIRT With Personalized Dosimetry
Brief Title: Pathological Results of Aggressive Hepatocellular Carcinomas Treated Using SIRT
Acronym: PAHCHS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0557
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to analyze pathological analysis of surgically treated aggressive hepatocellular carcinomas after radio-embolization.

The investigators aim to demonstrate that a higher dose results in better tumor response while respecting safety conditions, that is, no radiologically induced liver disease.

ELIGIBILITY:
Inclusion criteria:

- aggressive hepatocellular carcinomas with vascular invasion, large tumors or multifocal distribution

Exclusion criteria:

* Other treatment after SIRT (confounding effect)
* contraindications for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: aggressive hepatocellular carcinomas
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Pathological tumor response | 6 months
  Patients are treated with SIRT, then if the tumor response was adequate, surgery was performed.Analysis after surgery. (6 months after SIRT)

SECONDARY OUTCOMES:
Rate of Healthy liver hypertrophia | day 1
  Rate of Healthy liver hypertrophia

CONTACTS AND LOCATIONS:
Overall Officials: BORIS GUIU, PU-PH, Study Director — University Hospital, Montpellier; Mohamad MEERUN, intern, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Meerun MA, Allimant C, Riviere B, Herrero A, Panaro F, Assenat E, Cassinotto C, Mariano-Goulart D, Guiu B. Large, multifocal or portal vein-invading hepatocellular carcinoma (HCC) downstaged by Y90 using personalized dosimetry: safety, pathological results and outcomes after surgery. Hepatobiliary Surg Nutr. 2023 Jun 1;12(3):351-365. doi: 10.21037/hbsn-22-184. Epub 2022 Oct 31. PMID 37351147